CLINICAL TRIAL: NCT00599378
Title: Implementation Intentions to Promote Colon Cancer Screening in Rural Primary Care Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kimberly Engelman, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Kimberly Engelman, PhD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11018; 1R01CA121016-01A2 (NIH)
Record Dates: First submitted 2007-12-31; First posted 2008-01-23 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Implementation Intentions-based telephone counseling. Partnership intervention between rural Primary Care Physicians, their patients, and CRC Information Specialists using an implementation intentions based approach.
  Interventions: Behavioral: Implementation Intentions-based telephone counseling
- 2 (No Intervention): Healthy Living information on Physical Activity and Nutrition

INTERVENTIONS:
Behavioral: Implementation Intentions-based telephone counseling — Implementation Intentions-based telephone counseling
  Arms: 1

SUMMARY:
To assess the efficacy of a novel prompting intervention based on the concept of "implementation intentions.

DETAILED DESCRIPTION:
Although colorectal cancer (CRC) is preventable and curable if detected early, a large portion of the population is not current with screening recommendations. Many unscreened individuals 50 years of age and older do not receive health care system prompts to promote adherence to test preparation or completion. This study will assess the efficacy of a novel prompting intervention based on the concept of "implementation intentions". The intervention will be delivered through a partnership between patients, rural primary care physicians, and trained CRC information specialists (CRC-IS) and will focus on the 'recalcitrant' primary care population. A randomized design will test a comparison condition of a "no-partnership" system with generic information versus a "partnership" intervention system that specifically addresses each participants' CRC screening "implementation intentions" (the "when," "where" and "how" screening details). The study will be conducted with 600 patients eligible for CRC screening and recruited while presenting for care in a set of Research Network affiliated primary care clinics, or patient contact information gathered from in-house chart reviews. All participants who are not up-to-date on CRC screening, or not at high risk for CRC, will receive a baseline tablet PC-administered CRC assessment, or a letter of invitation from their PC physician to go online to the Healthy Living Kansas patient portal to complete the assessment. Completion of CRC screening at 60 days post index visit will be assessed through follow-up phone calls. Those not completing CRC screening after taking the assessment,(i.e., recalcitrant participants) then will be randomized to either C (comparison group-"no-partnership") or CPI2 (active intervention-CRC-IS/ physician/patient partnership and implementation intentions-based communication concepts). Physicians will receive informational fax sheets summarizing all participant phone calls. A 120-day post randomization follow-up telephone call will assess the effects of implementation intentions communications and perceived CRC screening barriers encountered. The primary outcome will be CRC screening adherence at 120 days. Secondary outcomes will assess 120-day perceived barriers and advancement in screening decisional stage. This intervention will provide information on the utility of embedding an "implementation intentions" based behavioral intervention for promoting CRC screening among initially non-adherent primary care patients.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* at average risk for colorectal cancer
* not up to date with colorectal cancer screening

Exclusion Criteria:

* Younger than 50 years of age
* at high risk for colorectal cancer
* up to date with colorectal cancer screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Follow up survey to assess participant compliance with CRC screening. For those non compliant participants, randomized to either Control group or CPI2 group - active intervention with implementation intentions-based communication concepts | 60 days

SECONDARY OUTCOMES:
120 day followup survey to assess perceived barriers and screening decisional stage | 120 Days

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly K. Engelman, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States